CLINICAL TRIAL: NCT01854970
Title: Benefit of Pharyngeal and Oesophageal pH-impedance of Patients With High Suspicion of Laryngopharyngeal Reflux
Acronym: PHARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2012/08
Record Dates: First submitted 2013-05-03; First posted 2013-05-16 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Laryngopharyngeal Reflux; Oesophageal pH-impedance
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Experimental)
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: esomeprazole — Patients with pharyngolaryngeal symptoms will have a clinical evaluation, laryngoscopy, and pharyngoesophageal pH-impedance. Then a treatment by esomeprazole during 8 weeks in the term of which the second clinical evaluation and pH-impedance will be made.

SUMMARY:
Laryngopharyngeal reflux (LPR) is the retrograde movement of gastric contents into the larynx, pharynx and upper aerodigestive tract. The symptoms and manifestations are very changeable and non specific. Pharyngeal and Oesophageal pH-impedance may help to detect these reflux and to identify patients with abnormal LPR.

To compare and describe the results of pharyngeal and oesophageal pH-impedance of patients with high suspicion of laryngopharyngeal reflux, with the results of healthy patients.

DETAILED DESCRIPTION:
This is a monocentric, prospective descriptive study. Patients will be recruited in otolaryngology and gastroenterology departments of Bordeaux teaching hospital. A first clinical, endoscopic and pH-impedance evaluation will be made, after at least 15 days of interruption of any proton pump inhibitors (PPI). After 8 weeks' treatment by double PPI doses (esomeprazole 40 mg bid), another clinical and pH-impedance evaluation will be realized. The characteristics of the patients who respond to the treatment will be compared to non responders. The subjects will also have an initial laryngoscopy, an oesophageal manometry allowing the location of the lower sphincter of the oesophagus and the upper sphincter of the oesophagus for positioning the catheters.

ELIGIBILITY:
Inclusion Criteria:

* age : 18 to 80 years old.
* Written consent
* Laryngopharyngeal symptoms (dysphonia, and/or globus and/or sensation, and/or pharyngeal pain, and/or cough) for 3 months at least.
* No PPI for at least 15 days
* Social security affiliation

Exclusion Criteria:

* Sinusitis or chronic rhinitis (in the previous year)
* Laryngeal trauma, tracheotomy or pharyngolaryngeal surgery
* pregnancy or absence of efficacy contraception
* breast feeding
* history of gastrointestinal pathology, diabetes, neurological condition
* cardio-vascular history requiring the taking of Plavix
* esomeprazole contraindication or intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of pharyngeal reflux/24h | visit 3 - 60 days after inclusion
• Number of pharyngeal acid reflux/24h | Visit 3 - 60 days after inclusion
• Number of pharyngeal less acid reflux/24h | Visit 3 - 60 days after inclusion
• Pharyngeal acid exposure (% of total time with pharyngeal pH <4) | Visit 3 - 60 days after inclusion
• Pharyngeal bolus exposure (% of total time with liquid in the pharynx) | Visit 3 - 60 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France